CLINICAL TRIAL: NCT01053091
Title: Effect of Exercise-based Rehabilitation on Circulatory Functions in Patients With Diastolic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Fu Tieh Cheng, attending physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98-1374B
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Heart Failure
Keywords: exercise-base rehabilitation; diastolic heart failure; cardiovascular function; aerobic fitness
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): exercise
  Interventions: Behavioral: exercise
- Control (No Intervention): control

INTERVENTIONS:
Behavioral: exercise — The trained subjects will be trained on a bicycle ergometer at about 60-70%of heart rate reserve for 35-55 minutes (that will include 10-min warm-up, 15-35-min main exercise, and 10-min cool-down) per day, 3 days per week for 12 weeks
  Other Names: behavioral
  Arms: Exercise

SUMMARY:
The purpose of this study is to investigate how exercise-base rehabilitation influences circulatory functions in patients with diastolic heart failure (DHF).

DETAILED DESCRIPTION:
A quasi-experimental design will be used in this investigation. Eighty DHF patients will be recruited from Chang Gung Medical Foundation, Keelung Branch after they have provided informed consent. These subjects will be randomized into the trained (n=40) and the control groups (n=40). The trained subjects will be trained on a bicycle ergometer at about 60-70%of heart rate reserve for 35-55 minutes (that will include 10-min warm-up, 15-35-min main exercise, and 10-min cool-down) per day, 3 days per week for 12 weeks. The control subjects will maintain their normal living pattern. Subjects' physical fitness, oxygen transport and utilization of exercising skeletal muscles, cardiovascular functions and hemodynamics, blood cell parameters, RBC deformity and aggregation, plasma biomarkers of myocardial damage, and thrombotic factors/reactions will be measured at pre-training stage and following the 8th and 12th week of the training program. Experimental results were analyzed by descriptive statistics (percentage, mean, and standard deviation), independent t-test, two-way ANOVA, and two-way ANCOVA. Previous researches were mainly focus on systolic heart failure, less on diastolic heart failure. We study the above parameter to realize the physiological response to exercise of these patients and discover the appropriate exercise intensity for prescription.

ELIGIBILITY:
Inclusion Criteria:

* cardiac event with optimal medial treatment within 3 months and have 4 more weeks spared from heart disease attack or major cardiac procedure.
* LVEF>50%

Exclusion Criteria:

* unstable angina pectoris,
* uncompensated heart failure,
* myocardial infarction during the past 4 weeks,
* complex ventricular arrhythmias,
* orthopedic or neurological limitations to exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
physical fitness including cardiovascular functions, oxygen transport and utilization of exercising skeletal muscles and hemodynamics | one year

SECONDARY OUTCOMES:
blood cell parameters, RBC deformity and aggregation, plasma biomarkers of myocardial damage, and thrombotic factors/reactions change between pre-ex and post-ex. | one year

CONTACTS AND LOCATIONS:
Overall Officials: T'sang-T'ang Hsieh, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation of Keelung Chang Gung Memorial hospital, Keelung, Taiwan

REFERENCES:
- [Background] Paulus WJ, Tschope C, Sanderson JE, Rusconi C, Flachskampf FA, Rademakers FE, Marino P, Smiseth OA, De Keulenaer G, Leite-Moreira AF, Borbely A, Edes I, Handoko ML, Heymans S, Pezzali N, Pieske B, Dickstein K, Fraser AG, Brutsaert DL. How to diagnose diastolic heart failure: a consensus statement on the diagnosis of heart failure with normal left ventricular ejection fraction by the Heart Failure and Echocardiography Associations of the European Society of Cardiology. Eur Heart J. 2007 Oct;28(20):2539-50. doi: 10.1093/eurheartj/ehm037. Epub 2007 Apr 11. PMID 17428822
- [Background] Loimaala A, Groundstroem K, Rinne M, Nenonen A, Huhtala H, Vuori I. Exercise training does not improve myocardial diastolic tissue velocities in Type 2 diabetes. Cardiovasc Ultrasound. 2007 Sep 26;5:32. doi: 10.1186/1476-7120-5-32. PMID 17897465
- [Background] Hunt SA, Abraham WT, Chin MH, Feldman AM, Francis GS, Ganiats TG, Jessup M, Konstam MA, Mancini DM, Michl K, Oates JA, Rahko PS, Silver MA, Stevenson LW, Yancy CW. 2009 focused update incorporated into the ACC/AHA 2005 Guidelines for the Diagnosis and Management of Heart Failure in Adults: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines: developed in collaboration with the International Society for Heart and Lung Transplantation. Circulation. 2009 Apr 14;119(14):e391-479. doi: 10.1161/CIRCULATIONAHA.109.192065. Epub 2009 Mar 26. No abstract available. PMID 19324966
- [Background] O'Connor CM, Whellan DJ, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Miller NH, Fleg JL, Schulman KA, McKelvie RS, Zannad F, Pina IL; HF-ACTION Investigators. Efficacy and safety of exercise training in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1439-50. doi: 10.1001/jama.2009.454. PMID 19351941
- [Background] Guazzi M, Myers J, Arena R. Cardiopulmonary exercise testing in the clinical and prognostic assessment of diastolic heart failure. J Am Coll Cardiol. 2005 Nov 15;46(10):1883-90. doi: 10.1016/j.jacc.2005.07.051. Epub 2005 Oct 24. PMID 16286176
- [Background] Maeder MT, Kaye DM. Heart failure with normal left ventricular ejection fraction. J Am Coll Cardiol. 2009 Mar 17;53(11):905-18. doi: 10.1016/j.jacc.2008.12.007. PMID 19281919
- [Derived] Fu TC, Yang NI, Wang CH, Cherng WJ, Chou SL, Pan TL, Wang JS. Aerobic Interval Training Elicits Different Hemodynamic Adaptations Between Heart Failure Patients with Preserved and Reduced Ejection Fraction. Am J Phys Med Rehabil. 2016 Jan;95(1):15-27. doi: 10.1097/PHM.0000000000000312. PMID 26053189